CLINICAL TRIAL: NCT02412163
Title: A Multicenter Study of Patients Treated With the Ellipse Technologies Intramedullary High Tibial Osteotomy (IM HTO) Nail System for Osteoarthritis and Varus Malalignment of the Knee
Brief Title: Ellipse Intramedullary Nail High Tibial Osteotomy Study
Acronym: IM HTO
Status: Completed | Type: Observational
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR0123
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Varus Malalignment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- IM HTO Nail: Implant with the Ellipse IM HTO Nail
  Interventions: Device: Ellipse IM HTO Nail

INTERVENTIONS:
Device: Ellipse IM HTO Nail

SUMMARY:
This study further evaluates the safety profile and efficacy of the Ellipse IM HTO Nail system in subjects with osteoarthritis and varus malalignment of the knee. All subjects will receive treatment with the Ellipse IM HTO Nail System and followed for six months.

DETAILED DESCRIPTION:
The Ellipse IM HTO Nail is intended for open wedge proximal tibial osteotomies. The Ellipse IM HTO Nail is an intramedullary nail that operates on the principles of distraction osteogenesis.

The Ellipse IM HTO Nail is used in valgizing HTO procedures to correct varus malalignment. The Ellipse IM HTO Nail is surgically placed in the intramedullary canal of the tibia. It is lengthened telescopically using the non-invasive external remote control.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has standing varus malalignment benefitting from high tibial osteotomy correction
2. Patient is diagnosed with current osteoarthritis of the knee
3. Patient is eighteen years of age or greater
4. Patient is a candidate to be implanted with an Ellipse IM HTO System
5. If female of childbearing potential, patient presents with a negative pregnancy test and agrees to employ adequate birth control measures for the duration of the study
6. Patient understands and accepts the obligation to comply with the required follow-up visits and is logistically able to meet all study requirements
7. Patient signs informed consent for the use of their personal private data

Exclusion Criteria:

1. Patient declines to sign informed consent for the use of their personal private data
2. Varus deformity greater than 10°
3. Flexion contracture greater than 15°
4. Knee flexion under 90°
5. Medial/lateral tibial subluxation over 1 cm
6. Medial bone loss of over 3 mm
7. Inflammatory arthritis
8. Arthritis in the lateral compartment
9. Patella baja
10. Weight over 114 kg
11. Severe patellofemoral symptoms
12. Unaddressed ligamentous instability
13. Fixed flexion contracture
14. Known or suspected osteoporosis or osteopenia based on medical history and radiographic images
15. Current use of nicotine products.
16. Requires other surgical procedures at the time of the HTO surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who meet the protocol eligibility criteria including standing varus malalignment in the limb presenting with osteoarthritis of the knee.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Weight-Bearing Line at Final Correction within ±5, 10, and 15% of Baseline Target | Pre-Op, Week 6 (Considered the Final Correction Visit unless additional visits are required)

SECONDARY OUTCOMES:
Absolute Difference in Weight-Bearing Line Final Target versus Actual at Final Consolidation | Week 6 (Considered the Final Correction Visit unless additional visits are required), Month 6 (Considered the Final Consolidation Visit unless additional visits are required)
Absolute Difference in Weight-Bearing Line Baseline Target versus Final Target | Pre-Op, Month 6 (Considered the Final Consolidation Visit unless additional visits are required)
  Baseline Target versus Final Target
Change in Hip-Knee-Ankle Angle Baseline versus Final Correction | Pre-Op, Week 6 (Considered the Final Correction Visit unless additional visits are required)
  Baseline versus Final Correction
Change in Hip-Knee-Ankle Angle Baseline versus Final Consolidation | Pre-Op, Month 6 (Considered the Final Consolidation Visit unless additional visits are required)
Change in Tibial Slope Angle Baseline versus Final Correction | Pre-Op, Week 6 (Considered the Final Correction Visit unless additional visits are required)
  Baseline versus Final Correction
Change in Tibial Slope Angle Baseline versus Final Consolidation | Pre-Op, Month 6 (Considered the Final Consolidation Visit unless additional visits are required)
  Baseline versus Final Consolidation
Time to Full Weight-Bearing | Week 2, Week 4, Week 6, Month 3, Month 6
  Amount of time required until a patient is allowed to put 100% of their body weight on the leg.

OTHER OUTCOMES:
Serious Adverse Events | Pre-Op, Operative, Week 2, Week 4, Week 6, Month 3, Month 6
  Incidence of Serious Adverse Events upon enrollment into the study
Unanticipated Adverse Device Effects | Pre-Op, Operative, Week 2, Week 4, Week 6, Month 3, Month 6
  Incidence of Unanticipated Adverse Effects upon enrollment into the study
Non-Serious Adverse Events | Pre-Op, Operative, Week 2, Week 4, Week 6, Month 3, Month 6
  Incidence of Non-Serious Adverse Events upon enrollment into the study
Secondary Surgical Procedures | Pre-Op, Operative, Week 2, Week 4, Week 6, Month 3, Month 6
  Incidence of Secondary Surgical Procedures upon enrollment into the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Dahl, MD, Principal Investigator — University of Minnesota
Locations (11):
- Medizinische Hochschule, Hanover, Germany
- Netherlands (2):
  - Martini Ziekenhuis, Groningen
  - Isala Klinieken, Zwolle
- Poland (4):
  - Centrum Ortopedii I Traumatologii, Bialystok
  - Zagiel Hospital, Lublin
  - Lekmed Hospital, Warsaw
  - District Hospital of Wolomin, Wołomin
- United Kingdom (4):
  - North Bristol NHS Trust, Bristol
  - North Cumbria University Hospital, Carlisle
  - University Hospital Aintree, Liverpool
  - University Hospitals Southampton, Southampton